CLINICAL TRIAL: NCT07133308
Title: A Double-Blind, Randomized, Placebo-Controlled Multicenter Study to Evaluate the Efficacy and Safety of Deuruxolitinib in Adolescent Patients With Severe Alopecia Areata With an Open-label Extension Period
Brief Title: Study to Evaluate the Efficacy and Safety of Deuruxolitinib in Adolescents With Severe Alopecia Areata
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Organization: Sun Pharmaceutical Industries Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP543.3101
Record Dates: First submitted 2025-07-29; First posted 2025-08-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: Treatment period:
  Model- Parallel Assignment, Number of Arms- 2
  The Treatment period will be followed by the Open-Label Extension Period:
  Model- Single Group Assignment, Number of Arms- 1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study subjects, Investigators, and site study staff will be blinded to study [Treatment Period] followed by None [Open-Label Extension]
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Period: Deuruxolitinib 8 mg (Experimental): Deuruxolitinib tablets, orally, twice daily (BID) for up to 24 weeks
  Interventions: Drug: Deuruxolitinib
- Treatment Period: Placebo (Placebo Comparator): Deuruxolitinib-matched placebo tablets, orally, BID for up to 24 weeks
  Interventions: Drug: Placebo
- Open-Label Extension: Deuruxolitinib 8 mg BID (Experimental): Deuruxolitinib tablets, orally, BID for up to 52 weeks
  Interventions: Drug: Deuruxolitinib

INTERVENTIONS:
Drug: Deuruxolitinib — Deuruxolitinib will be dosed orally as tablets at a dose of 8 mg
  Arms: Open-Label Extension: Deuruxolitinib 8 mg BID; Treatment Period: Deuruxolitinib 8 mg
Drug: Placebo — Deuruxolitinib matching placebo will be dosed orally as tablets
  Arms: Treatment Period: Placebo

SUMMARY:
This study evaluates the safety and effectiveness of deuruxolitinib in adolescents aged 12 to less than 18 years who have 50% or greater scalp hair loss.

DETAILED DESCRIPTION:
The efficacy and safety of deuruxolitinib in adolescent subjects with severe alopecia areata will be evaluated in this study, beginning with a double-blind, randomized, placebo-controlled Treatment Period of 24 weeks. Subjects 12 to <18 years of age having at least 50% hair loss as measured by SALT and meeting eligibility criteria will be randomized to deuruxolitinib or placebo treatment. In the Open-label Extension part of the study, participants from the Treatment Period will receive deuruxolitinib for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation compatible with alopecia areata with a current episode lasting at least 6 months and not exceeding 10 years.
* Between 12 to <18 years of age
* At least 50% scalp hair loss, as defined by a Severity of Alopecia Tool (SALT) score ≥50.
* Willing to comply with the study visits and requirements of the study protocol

Exclusion Criteria:

* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or other scalp condition that may interfere with the SALT assessment, or untreated actinic keratosis at Screening and/or Baseline
* Treatment with other medications or agents within 28 days of Baseline or during the study that may affect hair regrowth or immune response.
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug.
* Clinically significant medical condition, psychiatric disease, or social condition, as determined by the Investigator, that may unfavorably alter the risk-benefit of study participation, adversely affect study compliance, or confound interpretation of study results.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 355 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving an absolute Severity of Alopecia Tool (SALT) score ≤20 | Week 24
  SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).
Safety and tolerability of deuruxolitinib will be assessed by evaluating adverse events, vital signs, electrocardiograms, and clinical laboratory results, as well as physical examinations | Week 24
  Summary of participants who experience Treatment emergent adverse events (TEAEs) and serious TEAEs will be provided. An AE is defined as any untoward medical occurrence that may appear or worsen in a subject during the course of a study. Adverse events will be considered treatment-emergent if the onset is after the first dose of study drug. Summaries will be provided of participants who experience potentially clinically significant post-baseline changes in: hematology, chemistry and lipid results, vital signs (blood pressure, pulse rate, respiratory rate, temperature), electrocardiogram parameters (heart rate, PR, QT, QTcF, QRS, and RR) and physical examination findings.

SECONDARY OUTCOMES:
Percentage of subjects achieving an absolute SALT score of ≤20 | Weeks 4, 8, 12, 16, and 20
  SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).
Mean percent change (ie, relative change) in SALT scores from baseline | Weeks 4, 8, 12, 16, 20, and 24
  SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).
Percentage of responders (defined as "much improved" or "very much improved") using the Clinical Global Impression of Improvement (CGI-I) | Weeks 12, 16, 20, and 24
  The CGI-I is a questionnaire that asks the clinician to evaluate the improvement or worsening of the participant's alopecia areata as compared to the start of the study on a 7-point scale. Responses range from 1 (very much worse) to 7 (very much improved). Responders will defined as participants with responses of 6 (much improved) or 7 (very much improved).
Percentage of responders (defined as "much improved" or "very much improved") using the Patient Global Impression of Improvement (PGI-I) | Weeks 12, 16, 20, and 24
  The PGI-I is a self-administered questionnaire that asks the participant to evaluate the improvement or worsening of their alopecia areata as compared to the start of the study on a 7-point scale. Responses range from 1 (very much worse) to 7 (very much improved). Responders will be defined as participants with responses of 6 (much improved) or 7 (very much improved).
Mean change from baseline in the Clinical Global Impression of Severity (CGI-S) | Weeks 12, 16, 20, and 24
  The CGI-S is a questionnaire that asks the clinician to evaluate the symptom severity of the participant's alopecia areata at the time of assessment. The symptom severity was rated on a scale ranging from 1 to 7, where 1=normal, no hair loss; 2=borderline hair loss; 3=mild hair loss; 4=moderate hair loss; 5=marked hair loss; 6=severe hair loss; 7=among the most extreme hair loss. Higher scores indicate more hair loss. A negative change from baseline indicates less hair loss.
Mean change from baseline in the Patient Global Impression of Severity (PGI-S) | Weeks 12, 16, 20, and 24
  The PGI-S is a self-administered questionnaire that asks the participant to evaluate the symptom severity of their alopecia areata at the time of assessment. Symptom severity was rated on a scale ranging from 1 to 7, where 1=normal, no hair loss; 2=borderline hair loss; 3=mild hair loss; 4=moderate hair loss; 5=marked hair loss; 6=severe hair loss; 7=among the most extreme hair loss. Higher scores indicate more hair loss. A negative change from baseline indicates less hair loss.
Percentage of subjects achieving an absolute SALT score of ≤10 | Weeks 4, 8, 12, 16, 20, and 24
  SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).
Mean change from baseline on the Eyebrow Clinician-Reported Outcome (ClinRO) score | Weeks 4, 8, 12, 16, 20, and 24
  The Clinician-Reported Outcome Measure of Eyebrow Hair is a clinician-rated scale that assesses the total eyebrow hair present, based on a 4-point scale.
Mean change from baseline on the Eyelash Clinician-Reported Outcome (ClinRO) score | Weeks 4, 8, 12, 16, 20, and 24
  The Clinician-Reported Outcome Measure of Eyelash Hair is a clinician-rated scale that assesses the total eyelash hair present, based on a 4-point scale
Percentage of responders (defined as "satisfied" or "very satisfied") on the Satisfaction of Hair Patient Reported Outcome (SPRO) scale | Weeks 4, 8, 12, 16, 20, and 24
  SPRO is a questionnaire answered by the participant and designed to measure how satisfied alopecia areata participants are with their hair at the time of the assessment. The responses range from 1 to 5: 1= very satisfied, 2= satisfied, 3= neither satisfied nor dissatisfied, 4= dissatisfied, and 5= very dissatisfied. Higher scores indicate the greater hair dissatisfaction.
Mean change from baseline in the SPRO scale | Weeks 4, 8, 12, 16, 20, and 24
  SPRO is a questionnaire answered by the participant and designed to measure how satisfied alopecia areata participants are with their hair at the time of the assessment. The responses range from 1 to 5: 1= very satisfied, 2= satisfied, 3= neither satisfied nor dissatisfied, 4= dissatisfied, and 5= very dissatisfied. Higher scores indicate the greater hair dissatisfaction. A negative change from baseline indicate the greater hair satisfaction.
Percentage of subjects achieving SALT score of ≤ 20 at Week 24 whose SPRO rating shifted from Very Dissatisfied or Dissatisfied to Very Satisfied or Satisfied | Week 24
Percentage of subjects achieving SALT score of ≤ 10 at Week 24 whose SPRO rating shifted from Very dissatisfied or Dissatisfied to Very Satisfied or Satisfied | Week 24
Mean change from baseline on the individual items of the Quality of Hair Patient Reported Outcome (QPRO) scale | Weeks 4, 8, 12, 16, 20 and 24
  The QPRO questionnaire provides additional details on key attributes of hair and helps provide context to the SPRO response. The individual items of QPRO are: Satisfied thickness hair coverage; Satisfied evenness hair coverage; How satisfied with your eyebrows; How satisfied with your eyelashes, scored on a scale ranging from 1 to 5 where 1=very satisfied, 2=satisfied, 3=neither satisfied nor dissatisfied, 4=dissatisfied, 5=very dissatisfied. Higher scores indicate the greater dissatisfaction on hair quality. A negative change from baseline indicate the greater satisfaction on hair quality.
Mean change from baseline in total score of the Hospital Anxiety and Depression Scale (HADS) | Weeks 12 and 24
  HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Mean change from baseline in the depression scale of the HADS | Weeks 12 and 24
  HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Mean change from baseline in the anxiety scale of the HADS | Weeks 12 and 24
  HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Percentage of subjects achieving a ≥ 6-point change from baseline in total score of the HADS | Weeks 12 and 24
  HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Percentage of subjects achieving a ≥ 3-point change from baseline in the depression scale of the HADS | Weeks 12 and 24
  HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Percentage of subjects achieving a ≥ 4-point change from baseline in the anxiety scale in total score of the HADS | Weeks 12 and 24
  HADS is a questionnaire designed to assess anxiety and depression symptoms which is completed by participants. The questionnaire is comprised of two separate scales with a total of 14 items: A 7-item scale related to anxiety and 7-item scale related to depression. Each item within both scales is scored using a 4-point scale, ranging from 0 to 3 and the total scores in each scale can range from 0 to 21. Separate scores were created for anxiety and depression. A score between 0-7 is considered normal, 8-10 is mild, 11-14 is moderate, and >14 is severe anxiety or depression. Higher scores indicate greater severity. A negative change from baseline indicates less severity.
Proportion of Participants with Suicidal Ideation or Behavior Per the Columbia-Suicide Severity Rating Scale (C-SSRS) | Week 24
  C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions. Suicidal ideation is defined as a "yes" answer to either Questions 4 or 5 on the suicidal ideation section (with intent or plan).
Safety and tolerability of deuruxolitinib will be assessed by evaluating adverse events, vital signs, electrocardiograms, and clinical laboratory results, as well as physical examinations | Up to Week 80
  Summary of participants who experience Treatment emergent adverse events (TEAEs) and serious TEAEs will be provided. An AE is defined as any untoward medical occurrence that may appear or worsen in a subject during the course of a study. Adverse events will be considered treatment-emergent if the onset is after the first dose of study drug. Summaries will be provided of participants who experience potentially clinically significant post-baseline changes in: hematology, chemistry and lipid results, vital signs (blood pressure, pulse rate, respiratory rate, temperature), electrocardiogram parameters (heart rate, PR, QT, QTcF, QRS, and RR) and physical examination findings.
Effect of deuruxolitinib on treating Hair Loss as Measured by the Severity of Alopecia Tool (SALT) | Up to Week 76

CONTACTS AND LOCATIONS:
Locations (64):
- United States (54):
  - Total Skin And Beauty Dermatology Center, Birmingham, Alabama
  - Avacare - Cct Research - Center For Dermatology And Plastic Surgery, Scottsdale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Kern Research Inc., Bakersfield, California
  - Center For Dermatology Clinical Research Inc., Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Palmtree Clinical Research, Palm Springs, California
  - Paradigm Clinical Research - San Diego, San Diego, California
  - Colorado Medical Research Center, Denver, Colorado
  - Paradigm Clinical Research - Wheat Ridge, Wheat Ridge, Colorado
  - D&H Doral Research Center, Doral, Florida
  - Skin Care Research, Llc - Hollywood, Hollywood, Florida
  - Ilumina Medical Research Llc, Kissimmee, Florida
  - All X Ray Diagnostic Services Corp, Miami, Florida
  - Millennium Medical Research Llc, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - Florida Pharmaceutical Research And Associates, Inc., Miami, Florida
  - L&C Professional Medical Research Institute, Miami, Florida
  - Pediatric Skin Research Llc, Miami, Florida
  - Valencia Medical & Research Center, Miami, Florida
  - Advance Research Center, Llc, Miami, Florida
  - Barroso Medical Services Llc, Miami Lakes, Florida
  - Nexus Research Llc, Pompano Beach, Florida
  - International Clinical Research Us Llc - Sanford, Sanford, Florida
  - Lenus Research & Medical Group Llc., Sweetwater, Florida
  - Cleaver Medical Group Dermatology, Cumming, Georgia
  - Skin Care Physicians Of Georgia, Macon, Georgia
  - Georgia Skin & Cancer Clinic, Savannah, Georgia
  - Asr, Llc, Boise, Idaho
  - Denova Research, Chicago, Illinois
  - Ds Research - Indiana, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group Llc., Indianapolis, Indiana
  - Ds Research - Kentucky, Louisville, Kentucky
  - U.S. Dermatology Partners - Rockville, Rockville, Maryland
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Revival Research Institute, Llc - Troy, Mi, Troy, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Boeson Research Mso, Missoula, Montana
  - Skin Specialists, Pc, Omaha, Nebraska
  - Schweiger Dermatology & Allergy - Verona, Verona, New Jersey
  - Vitality Clinical Trials, Woodbury, New York
  - Revival Research Institute, Llc - Cary, Nc, Cary, North Carolina
  - Darst Dermatology, Charlotte, North Carolina
  - Dermatologists Of Southwest Ohio, Mason, Ohio
  - Dermatology Associates Of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Tribe Clinical Research, Llc, Greenville, South Carolina
  - Delricht Research - Smyrna, Smyrna, Tennessee
  - Dermatology Treatment And Research Center - Dallas, Dallas, Texas
  - North Texas Center For Clinical Research, Frisco, Texas
  - Austin Institute For Clinical Research Inc., Pflugerville, Texas
  - Texas Dermatology And Laser Specialists, San Antonio, Texas
  - Jordan Valley Dermatology, South Jordan, Utah
  - Avacare - Cct Research - Springville Dermatology, Springville, Utah
  - National Eagle Research, Llc, Lynnwood, Washington
- Canada (10):
  - Kirk Barber Research, Calgary, Alberta
  - Dermatology Research Institute (Calgary), Calgary, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - Care Clinic Ltd., Red Deer, Alberta
  - Medical Arts Health Research Group - Kelowna, Kelowna, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Lynderm Research Inc., Markham, Ontario
  - Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario
  - Research Toronto, Toronto, Ontario
  - Facet Dermatology, Toronto